CLINICAL TRIAL: NCT01425125
Title: Study of Nonedematous Hyponatremia and the Utility of Fractional Urate Excretion in Hyponatremia and Suspected Renal Salt Wasting Without Hyponatremia-
Brief Title: Fractional Urate Excretion in Nonedematous Hyponatremia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10029; 10029 (Other: Winthrop University Hospital IRB)
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Cerebral Hyponatremia; SIADH; Cerebral Salt-wasting Syndrome; Reset Hypothalamic Osmostat
Keywords: nonedematous hyponatremia; fractional urate excretion
MeSH Terms: conditions — Inappropriate ADH Syndrome | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tolvaptan in euvolemic hyponatremia (Experimental): This arm will test the effectiveness of tolvaptan in treating the hyponatremia of patients with euvolemic hyponatremia.
  Interventions: Drug: Tolvaptan in euvolemic hyponatremia

INTERVENTIONS:
Drug: Tolvaptan in euvolemic hyponatremia — This arm will test the effectiveness of tolvaptan in treating the hyponatremia of patients with euvolemic hyponatremia.
  Other Names: oral tolvaptan (Samsca

SUMMARY:
Hyponatremia, defined as a serum sodium < 135 mmol/l, in patients without edema has undergone significant changes where it is now evident that even mild hyponatremia should be treated because of its association with symptoms, especially a fourfold increase in falls over the age of 65 years. There is an unresolved controversy over the relative prevalence of the syndrome of inappropriate secretion of antidiuretic hormone (SIADH) and cerebral/renal salt wasting (C/RSW). Resolution of this diagnostic dilemma becomes urgent because of divergent therapeutic goals, to water-restrict in SIADH or to give salt and water supplementation in C/RSW. The dilemma is compounded by recent reports of C/RSW occurring in patients without cerebral disease, thus adding further confusion in defining the relative prevalence of both syndromes. Because of overlapping laboratory and clinical findings in both syndromes, only differences in the state of extracellular volume differentiates one syndrome from the other, being high normal to increased in SIADH and decreased in C/RSW. The investigators have used fractional excretion (FE) of urate to categorize patients with hyponatremia. The increased FEurate that is observed in hyponatremic patients with SIADH and C/RSW can be used to differentiate both syndromes by correcting the hyponatremia and determining whether FEurate normalizes as in SIADH or remains increased in C/RSW. The present studies have been designed to determine total body water by deuterium and extracellular water by sodium bromide in patients with nonedematous hyponatremia with normal and increased FEurate to differentiate more conclusively whether the patient has normal or decreased water volumes. The investigators will also correct serum sodium rapidly with judicious administration of hypertonic saline over approximately three days and determine whether FEurate normalizes as in SIADH or remains increased as in C/RSW. In another group of patients, The investigators have data to suggest that those with normal sodium and increased FEurate is consistent with C/RSW. The investigators intend to do the same water volume studies to determine whether an increased FEurate with normonatremia would have decreased total and extracellular water that these patients have C/RSW without the need to correct a prior hyponatremia.

DETAILED DESCRIPTION:
The investigators have demonstrated that a normal FEurate in a nonedematous hyponatremic patient is highly consistent with the diagnosis of reset osmostat (RO). Since as much as 36% of patients with SIADH have RO, the investigators will evaluate these patients by either noting dilute urines in spontaneously excreted urines or after a modified water-loading test. The investigators have found that a normal FEurate in a nonedematous hyponatremic patient is highly consistent with RO.

The investigators intend to treat euvolemic patients with hyponatremia with tolvaptan, the V2 ADH receptor blocker, to determine the effectiveness of this form of therapy in a group of patients in whom correction of hyponatremia has been difficult to achieve by usual methods.

Nonedematous hyponatremic patients with serum sodium < 135 mmol/l will be recruited from Winthrop-University Hospital and from our outpatient practice.

It is anticipated that the present studies will provide valuable information on the relative prevalence of SIADH and C/RSW in patients with nonedematous hyponatremia. One possible drawback to these studies is our inability to determine total and extracellular water volumes in patient who are admitted to the neuro/neurosurgical ICU where the acute illnesses require parenteral therapy that will create a nonsteady state situation where total and extracellular water volumes cannot be accurately determined. This is an important possible omission because volume studies in this population of studies have indicated more that two thirds of patients having decreased volumes that were consistent with C/RSW, yet the medical literature states that C/RSW is rare. Studies in hyponatremics elsewhere in the hospital should shed important light on the methods to differentiate SIADH from C/RSW, data which can assist us in differentiating both syndromes in the neuro/neurosurgical ICU, where the investigators intend to perform FEurates.

It is anticipated that volume studies in patients with Alzheimer's disease with normal serum sodium and increased FEurate will demonstrated decreased volumes and confirm our earlier observations that many of these patients are renal salt wasters. It would be interesting to test whether volume repletion with saline will improve them mentally and physically.

ELIGIBILITY:
Inclusion Criteria:

- Nonedematous hyponatremia with normal renal, adrenal and thyroid function. -Non-hyponatremia with increased fractional excretion of urate.

Exclusion Criteria:

* Subjects < 18 years of age
* Pregnancy
* Serum creatinine > 1.4 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Etiologic categorization of nonedematous hyponatremia | 2 years
  We will attempt to categorize the etiology of nonedematous hyponatremia by the following parameters in decreasing order of importance, total and extracellular water determinations, fractional urate excretion, plasma renin and aldosterone levels, urinary sodium concentration and urine osmolality. We will also determine total and extracellular water in a group suspected of having renal salt wasting by virtue of having increased fractional urate excretion and normal serum sodium concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: John K Maesaka, MD, Principal Investigator — Winthrop University Hospital; Louis J Imbriano, MD, Study Director — Winthrop University Hospital
Locations (1):
- Winthrop-University Hospital, Mineola, New York, United States